CLINICAL TRIAL: NCT06028737
Title: Total Neoadjuvant Chemotherapy With 5-fluoruracil, Leucovorin, Oxaliplatin, and Docetaxel in Locally Advanced Gastric and Gastroesophageal Junction Cancer (OCTASUR): Randomized, Multi-center, Open-label Trial, Phase 2/3
Brief Title: Total Neoadjuvant FLOT Chemotherapy in Locally Advanced Gastric and Gastroesophageal Junction Cancer
Acronym: OCTASUR
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ukrainian Society of Clinical Oncology (Other)
Responsible Party: Principal Investigator, Mykyta Pepenin, MD, Ukrainian Society of Clinical Oncology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 241/4
Record Dates: First submitted 2023-08-26; First posted 2023-09-08 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Gastric Cancer; Stomach Cancer; GastroEsophageal Cancer; Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma; Advanced Gastric Adenocarcinoma; Gastric Neoplasm; Stomach Neoplasm; Gastrointestinal Cancer; Advanced Gastroesophageal Junction Adenocarcinoma; Advanced Gastric Carcinoma; Chemotherapy; Gastrectomy; Gastrectomy for Gastric Cancer; Gastric Resection; Gastric (Cardia, Body) Cancer
Keywords: Total neoadjuvant chemotherapy; FLOT; Fluoruracil; Gastrectomy; Perioperative chemotherapy; Docetaxel; Leucovorin; Gastric resection; Gastric cancer
MeSH Terms: conditions — Stomach Neoplasms; Gastrointestinal Neoplasms; Neoplasms | interventions — Docetaxel; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Perioperative 4+4 FLOT cycles (Active Comparator): 4 cycles of neoadjuvant FLOT chemotherapy regimen, followed by surgery and 4 cycles of adjuvant FLOT chemotherapy regimen.
  Interventions: Drug: Docetaxel; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Fluorouracil
- Total Neoadjuvant ChemoTherapy (TNT) 8 FLOT cycles (Experimental): 8 cycles of total neoadjuvant FLOT chemotherapy regimen, followed by surgery.
  Interventions: Drug: Docetaxel; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Fluorouracil

INTERVENTIONS:
Drug: Docetaxel — 50mg/m2, d1, i.v., every 2 weeks
Drug: Oxaliplatin — 85 mg/m², d1, i.v., every 2 weeks
Drug: Leucovorin — 200 mg/m², d1, i.v., every 2 weeks
Drug: Fluorouracil — 2600 mg/m²d1 i.v. every 2 weeks

SUMMARY:
The main goal of this study is to investigate the proportion of participants with locally advanced gastric and gastroesophageal adenocarcinoma without previous treatment during the last 5 years who can tolerate all planned cycles of chemotherapy and radical surgical treatment who will be prospectively randomized into two groups to undergo one of two chemotherapy regimens, followed by surgery:

1. 8 cycles of Total Neoadjuvant ChemoTherapy (TNT) with 5-Fluorouracil (5-FU), Leucovorin, Oxaliplatin, and Docetaxel (FLOT) followed by surgery.
2. 4 cycles of Neoadjuvant FLOT chemotherapy scheme preoperatively and 4 adjuvant FLOT cycles postoperatively.

DETAILED DESCRIPTION:
This is a multi-center international European prospective randomized study that aims to enroll participants with resectable locally advanced gastric and gastroesophageal (Siewert 2, 3) adenocarcinoma (≥cT3 and/or ≥cN0 and M0) with no history of previous oncological treatment during the last five years, who will be included in this study after reading and signing the informed consent. After the initial diagnostic laparoscopy, patients will be randomized into two groups in a 1:1 ratio, with allocation to one of the two study groups.

Patients randomized to the first (control) group will receive eight cycles of the perioperative FLOT chemotherapy scheme: 4 cycles before surgical treatment and four cycles after surgical intervention. Patients randomized to the second (study) group will receive eight cycles of FLOT total neoadjuvant chemotherapy, followed by surgery.

The study's primary endpoint is the proportion of patients receiving all planned chemotherapy cycles and radical surgical treatment. Secondary endpoints are perioperative morbidity and mortality (surgical and chemotherapeutic complications); disease-free survival (DFS) and 1-, 3- and 5-years overall survival (OS); quality of life during and after the treatment; correlation between the pathohistological response and chemotherapy regimen; composition and biomarkers of gut microbiota; objective tumor response.

Based on previous studies, with the current standard treatment protocol-four cycles of FLOT chemotherapy before surgery and four cycles after-only 47% of patients complete all eight cycles. In contrast, with total neoadjuvant therapy, where the entire chemotherapy regimen is administered before surgery, 71% of patients are able to complete all eight FLOT cycles.

Given these findings, it was calculated that to ensure 80% study power with a two-sided 5% significance level, each study group should include 65 participants. Considering an expected dropout rate of 15%, a total of 150 patients will be recruited. Up to 40 patients will be enrolled in Vilnius, Lithuania, with the remaining participants recruited in Kyiv, Ukraine.

ELIGIBILITY:
Inclusion Criteria:

* Tumor spread according to TNM: ≥cT3 and/or ≥cN0 and M0 (except of invasion of the common hepatic artery, celiac trunk, proximal part of the splenic artery, aorta, head of the pancreas);
* Performance status by Eastern Cooperative Oncology Group (ECOG): 0 - 1;
* Histologically confirmed gastric adenocarcinoma or gastroesophageal junction (Siewert type 2/3) adenocarcinoma.
* Differentiation grade: G0 - G4;
* Tumor localization: cardio-esophageal junction (Siewert 2, 3), cardiac part of the stomach, body of the stomach, antral part of the stomach, pyloric part of the stomach;
* Tumor extension: esophagus, diaphragm, liver, body and tail of the pancreas, anterior abdominal wall, small and large intestine, distal part of the splenic artery, spleen;
* Patient agrees to participate in this biomedical study.

Exclusion Criteria:

* Presence of another oncological disease at a different site if less than 5 years have passed since radical treatment.
* Comorbidities or patient conditions that preclude the administration of chemotherapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2027-04-25 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
All 8 planned FLOT cycles tolerance rate. | From enrollment to the end of treatment at 12 weeks
  The proportion of patients receiving all planned cycles of chemotherapy and radical surgical treatment.

SECONDARY OUTCOMES:
Chemotherapy toxicity rate and profile. | At the end of each FLOT cycle (each cycle is 14 days), up to 14 days after the last cycle.
  To determine chemotherapeutic toxicity profile, according to Common Terminology Criteria for Adverse Events (CTCEA 5.0).
Surgical complications rate. | 30 days after surgery.
  To determine postoperative surgical complications rate and profile after the different chemotherapy regimens, according to Clavien-Dindo classification.
Median overall survival. | From the start of treatment to the patient's death or the end of follow-up - 5 years follow-up after the last intervention.
  To determine the efficacy of TNT FLOT regimen compared to perioperative FLOT regimen by assessment of overall survival.
Progression-free survival. | Calculated as the time from the start of treatment to disease progression or the end of follow-up at 5 years after the treatment completion.
  To determine the efficacy of total neoadjuvant FLOT regimen compared to perioperative FLOT regimen.
Quality of patients' life. | 24 months.
  To determine the quality of life during the chemotherapy in both groups, after the surgery and 2 years follow-up after the treatment completion, assessed using a standardized European Organisation for Research and Treatment of Cancer quality-of-life questionnaire Core Questionnaire (EORTC QLQ-C30). Values from 30 to 126 mean a better or worse outcome, respectively.
Quality of patients' life. | 24 months.
  To determine the quality of life during the chemotherapy in both groups, after the surgery and 2 years follow-up after the completion of treatment, assessed using standardized European Organisation for Research and Treatment of Cancer quality-of-life questionnaires for Gastric Cancer (EORTC QLQ-STO22). Values from 22-88 mean a better or worse outcome, respectively.
Correlation between the pathohistological response and overall and disease-free survival. | 21 days after surgery.
  To determine the correlation between the pathohistological response and overall and progression-free survival, using the Becker criteria.
Histopathological tumor response rate (Becker regression criteria). | 21 days after surgery
  To determine the pathohistological regression rate after 8 FLOT cycles in total neoadjuvant regimen compared to 4 FLOT cycles in neoadjuvant regimen.
Intestinal microbiome composition. | Within 7 days before the start of the treatment.
  Significant differences in the alpha-diversity of the intestinal microbiome between patients with a good and poor response to neoadjuvant chemotherapy.
Objective tumor response. | From within 7 days before the first chemotherapy course and until 4 weeks before the surgical intervention.
  Assessed according to RECIST v1.1 criteria based on preoperative and control computed tomography.

CONTACTS AND LOCATIONS:
Overall Officials: Mykyta Pepenin, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- National Cancer Institute, Vilnius, Lithuania
- National Cancer Institute, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
After the initial publication every participant will receive all the data to provide further data exploration.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available after initial paper is published.